CLINICAL TRIAL: NCT04094493
Title: Role of Pre Operative Vit D Administiration in Decrease Incidence of Post Thyroidectomy Hypocalcemia
Brief Title: Vit D Role in Post Thyroidectomy Hypocalcemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ramadan, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: pre-thyroidectomy vit D
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Diseases
Keywords: thyroid - thyroidectomy - hypocalcemia - Vit D administiration
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 (Experimental): vit D + no hypocalcemia
  Interventions: Drug: vit D
- A2 (Experimental): Vit D + hypocalcemia
  Interventions: Drug: vit D
- B1 (No Intervention): NO vit D + no hypocalcemia
- B2 (No Intervention): NO vit D + hypocalcemia

INTERVENTIONS:
Drug: vit D — preoperative intra muscular vit D injection
  Arms: A1; A2

SUMMARY:
Hypocalcemia after total thyroidectomy is usually transient but it is of main concern as it requires either prolonged stay in the hospital or readmission. During the first 24 hours bleeding is the main complication, but from the second day to six months, transient hypocalcemia is of main concern. Hypocalcemia can be evaluated symptomatically as well as from laboratory testing. Signs and symptoms of hypocalcemia include numbness, tingling, and carpopedal spasm. Preoperative vitamin D prevents postoperative transient hypocalcemia after thyroidectomy .

DETAILED DESCRIPTION:
Thyroid surgery is one of the most frequently performed surgical procedures worldwide . Nowadays, total thyroidectomy is the recommended procedure for thyroid disease . As total thyroidectomy is the procedure of choice, the most common complication resulting after this surgery is transient hypocalcemia - the incidence being 24% - which increases the morbidity rate and increases the length of hospitalization . Other complications of thyroidectomy include recurrent laryngeal nerve injury which leads to hoarseness of voice, postoperative hemorrhage, dysphagia due to inflammation of the tissues surrounding the esophagus, seroma formation, Horner's syndrome due to injury to the cervical sympathetic chain, and poor healing of the wound with hypertrophy of the scar or wound infection .

Advances in surgical techniques have evolved to preserve the parathyroid gland function, which helps to prevent permanent hypocalcemia and its incidence now has reduced to 1-2% . However, transient hypoparathyroidism still occurs resulting in transient hypocalcemia. It occurs due to the age, parathyroid gland handling, devascularization, venous congestion, post-surgical local site edema and neck dissection . Prescribing preoperative vitamin D and calcium decreases the incidence of transient hypocalcemia after total thyroidectomy from 25.9% to 6.8% as compared to the control group .

Total thyroidectomy is the procedure of choice in our population with the preservation of the parathyroid gland. As transient hypocalcemia is common in post-thyroidectomy patients and increases the morbidity rate, giving vitamin D and calcium preoperatively can reduce the burden of postoperative transient hypocalcemia and it will be helpful in decreasing the morbidity rate due to post-thyroidectomy transient hypocalcemia. The objective of our study is to compare the frequency of transient hypocalcemia after vitamin D with the control group for patients undergoing total thyroidectomy.

The study is based on patients with thyroid diseases who are indicated for total thyroidectomy . Patients are divided into two groups : group A who will recieve Vit D before operation and group B who won't . Group A will be divided into :

A1 : no hypocacemia occurs with vit D A2 : hypocalcemia occurs with vit D .

Group B will be divided into:

B1 no hypocacemia without vit D B2 hypocalcemia without vit D . Comparison between the above mentioned four groups will determine the effectiveness of vit D in normalization of serum calcium levels after total thyroidectomy .

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patient age: > 18 years
* surgical indication for total thyroidectomy
* normal preoperative serum calcium level

Exclusion Criteria:

* Low preoperative calcium level
* Renal impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum calcium level | 2nd day post operatively
  normal serum calcium level above 8.8 is the target
Appearance of hypocalcemic tetany | 2nd day post operatively
  numbness , tingling or carpopedal spasm are undesirable clinical presentation of hypocalcemia

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khan Bhettani M, Rehman M, Ahmed M, Altaf HN, Choudry UK, Khan KH. Role of pre-operative vitamin D supplementation to reduce post-thyroidectomy hypocalcemia; Cohort study. Int J Surg. 2019 Nov;71:85-90. doi: 10.1016/j.ijsu.2019.08.035. Epub 2019 Sep 5. PMID 31494332
- [Result] Xing T, Hu Y, Wang B, Zhu J. Role of oral calcium supplementation alone or with vitamin D in preventing post-thyroidectomy hypocalcaemia: A meta-analysis. Medicine (Baltimore). 2019 Feb;98(8):e14455. doi: 10.1097/MD.0000000000014455. PMID 30813146
- [Result] Soares CSP, Tagliarini JV, Mazeto GMFS. Preoperative vitamin D level as a post-total thyroidectomy hypocalcemia predictor: a prospective study. Braz J Otorhinolaryngol. 2021 Jan-Feb;87(1):85-89. doi: 10.1016/j.bjorl.2019.07.001. Epub 2019 Aug 6. PMID 31492617
- [Result] Cherian AJ, Ponraj S, Gowri S M, Ramakant P, Paul TV, Abraham DT, Paul MJ. The role of vitamin D in post-thyroidectomy hypocalcemia: Still an enigma. Surgery. 2016 Feb;159(2):532-8. doi: 10.1016/j.surg.2015.08.014. Epub 2015 Sep 11. PMID 26365947
- [Result] Docimo G, Tolone S, Pasquali D, Conzo G, D'Alessandro A, Casalino G, Gili S, Brusciano L, Gubitosi A, Del Genio G, Ruggiero R, Docimo L. Role of pre and post-operative oral calcium and vitamin D supplements in prevention of hypocalcemia after total thyroidectomy. G Chir. 2012 Nov-Dec;33(11-12):374-8. PMID 23140919